CLINICAL TRIAL: NCT05629624
Title: Multidimensional Evaluation of the Early Emergence of Executive Function and Emotional Regulation in Young Children in Bangladesh Using Nutritional and Psychosocial Intervention: A Pilot Study
Brief Title: Evaluation of Executive Function and Emotional Regulation in Children in Bangladesh
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Boston Children's Hospital (Other)
Collaborators: The University of The West Indies (Other); International Centre for Diarrhoeal Disease Research, Bangladesh (Other); University of Auckland, New Zealand (Other); Wellcome Trust (Other)
Responsible Party: Principal Investigator, Charles Alexander Nelson III, Professor of Pediatrics and Neuroscience, Boston Children's Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: M4EFaD/Dhaka PR-21084
Record Dates: First submitted 2022-10-04; First posted 2022-11-29 (Actual); Last update posted 2022-11-29 (Actual); Status verified 2022-11

CONDITIONS: Executive Function Disorder; Emotional Regulation; Malnutrition, Child
Keywords: Executive Function; Emotional Regulation; Malnutrition; Children; Bangladesh
MeSH Terms: conditions — Emotional Regulation; Child Nutrition Disorders; Malnutrition

STUDY DESIGN:
Intervention Model Description: We will recruit a sample of malnourished children and randomly assign to different intervention arms. We will also have a control sample of well-nourished children for comparison analysis.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Chickpea based RUSF (Experimental): Locally produced ready to use supplementary food (RUSF), 50 g/packet contains 204 kcal energy). Two packets of RUSF provided for consumption at a rate of 50-100 kcal/kg/day till the child's weight for height returns to normal (WHZ >-1SD) or for maximum 3 months.
  Interventions: Dietary Supplement: Chickpea based RUSF
- E-RUSF (Experimental): Enhanced Ready to use therapeutic feeds (E-RUSF), 50-100 kcal/kg/d daily until for anthropometric recovery (WHZ > - 1SD) is achieved or for maximum 3 months then E-SQLNS will be given till the end of 2 years follow-up.
  Interventions: Dietary Supplement: E-RUSF
- Well-nourished children (No Intervention): Well-nourished children at 1 year of age (WLZ/WHZ score >-1 SD). No nutritional or psychosocial intervention. Only follow-up.
- Outcome reference group (Experimental): 3 year olds previously untreated MAM children (WHZ <-2 and ≥-3 z-score, and/or MUAC <12.5 and ≥11.5 cm) and free from any acute illness will be used as the outcome reference group.
  Interventions: Dietary Supplement: Outcome reference group/RUSF

INTERVENTIONS:
Dietary Supplement: Chickpea based RUSF — One group will receive locally produced RUSF, approximate at 50-100 kcal/kg/day, two of 50g packets daily (42) until anthropometric recovery ( WHZ > - 1SD) has been achieved or for maximum 3 months then immediately 1 packet / day SQLNS will be given throughout the study till the end of 2 years of follow-up.
  Arms: Chickpea based RUSF
Dietary Supplement: E-RUSF — The other group will receive the E-RUSF at 50-100 kcal/kg/day which in this age group approximates one 92 g sachet daily until anthropometric recovery ( WHZ > - 1SD) has been achieved or for a of maximum 3 months, then immediately E-SQLNS 1 packet daily provided throughout the study till the end of 2 years of follow-up.
  Arms: E-RUSF
Dietary Supplement: Outcome reference group/RUSF — We will also recruit 70 three-year-old previously untreated MAM children WHZ <-2 and ≥-3 z-score, and/or MUAC <12.5 and ≥11.5 cm as an outcome reference group for a singular assessment. All children (both case & control) will undergo a baseline nutritional, medical, biological and neuropsychological assessment (EF, ER, EEG and fNIRS). After all the assessments chick-pea based RUSF will be given for 2 months for nutritional rehabilitation.
  Arms: Outcome reference group

SUMMARY:
The study explores the impact of malnutrition at enrollment on executive function (EF) and emotional regulation (ER) in malnourished 1-year-old children and whether specially designed brain directed therapeutic feeds improve EF/ER outcomes at three years of age. The study will detect changes in EF and ER related to nutritional rehabilitation using specially designed ready to use therapeutic feeds (E-RUSF Nutriset) during the repletion phase and maintained for two years until age 3 with enhanced E-SQLNS (small quantity lipid based nutrient supplement) also modified to provide adequate brain directed micro and macronutrients. The investigators hypothesize that standard Bangladeshi designed B-RUSF and SQLNS (Nutriset) do not provide adequate nutrients to supply the brain during the rapid catch-up growth and subsequent early childhood growth phases of rehabilitation from Moderate Acute Malnutrition (MAM). The investigators predict that the children with moderately severe malnutrition treated with E-RUSF followed by 2 years of E-SQLNS will show an exuberance of connections (higher functional connectivity) than children receiving standard Bangladeshi rehabilitation feeds B-RUSF and SQLNS. This prediction is based on past work using EEG to examine the BEAN sample in Bangladesh, and differs from the sample in Boston, where the investigators anticipate that among healthy, normally nourished children, greater connectivity will be associated with better cognitive outcomes. The Core Toolkit will be deployed to the Bangladesh site to define its utility in prediction of executive dysfunction and emotional dysregulation in the context of low-income status, malnutrition and nutritional intervention. All nutritional intervention groups of malnourished children will also receive a set psychosocial stimulation curriculum that has been shown to be effective on severely malnourished children with therapeutic feedings.

DETAILED DESCRIPTION:
Malnutrition affects around 47 million children under 5 years of age annually and underlies 45% of the mortality in low- and middle-income countries where around 2 billion survivors suffer long term cognitive and behavioural sequelae. Acute malnutrition, comprising both MAM (Moderate Acute Malnutrition) and SAM (Severe Acute Malnutrition) causes 14.6% of all deaths of children under 5 years of age globally. It is a significant problem in Bangladesh where > 40% of under-fives have chronic or moderately acute malnutrition. The long-term consequences of malnutrition for the 5.5 million children under 5 years that suffer from chronic malnutrition (stunting or low height-for-age) and the 14% are acutely malnourished (wasting or low weight-for-height) include poor brain development with resultant impairment of the development of cognitive, motor, and socio-emotional skills throughout childhood and adulthood. Malnutrition during early childhood negatively affects cognition, behaviour, school performance and productivity in later life. Further, current rehabilitation feeding regimes do not reverse the impairment in brain development as these are designed with rapid catch-up growth as the principal goal.

Malnourished children have an abnormal assembly of the early gut microbiota which may impair brain function by disturbing the bidirectional neural and immune interactions between gut and brain by altered production of signal molecules by the microbiota such as short-chain fatty acids, and neurotransmitters. Nutritionally wasted children notably have marked brain atrophy on MRI and while re-feeding reverses brain atrophy, significant deficits remain in function and microstructure. It is likely that the anatomic reconstitution of the brain with feeds designed principally for corporal rapid catch-up growth results in brain structure which is unable to provide substrate for normal cognitive and emotional performance. Fixing this must depend at least in part on provision of the appropriate nutrients in amounts that meet demands during rapid catch-up growth of the body and brain.

The investigators propose that nutrient deficiencies, and gut microbiome dysbiosis both induce structural and functional abnormalities of the brain in malnutrition that lead to neuropsychological sequelae in childhood and later life. The human brain develops during intrauterine life as well as early childhood, especially in the developmental window between birth and 3 years of age. Better recovery of brain architecture and function in children suffering malnutrition will result from augmenting feeds with key nutrients with targeted functionality in the brain during rapid brain regrowth. The supplements are E-RUSF (Ready to Use Therapeutic Feed-enhanced manufactured by Nutriset) and E-SQLNS (standard/enhanced small quantity lipid based nutrient supplements) all containing key nutrients for rehabilitating wasted brains: 24 micronutrients (vitamins and minerals) provided at recommended daily allowance levels, functional lipids (Long Chain Polyunsaturated Fatty Acids DHA and EPA), sialylated milk oligosaccharides, neural specific antioxidants (zeaxanthine, lutein; crypto-xanthine) and microbiome modulating dietary soluble fibre mix (inulin + FOS), 6 g per 26g daily dose of E-SQLNS, as well as within a daily 100g ration of E-RUSF. The comparator group will receive standard of care therapeutic feeds in Bangladesh. These feeds are an energy dense chickpea-based RUSF with a targeted calorie delivery of 250 kcal/50 g (per serving) with caloric distribution 45-50 percent from fat and 8-10 percent from protein.

The diagnostic criteria for MAM in children 6 to 59 months of age are weight-for-height z-score <-2 and ≥-3 z-score of WHO child growth standards and/or MUAC <12.5 and ≥11.5 cm. This definition is also supported by USAID. There are about 1.8 million children under 5 years of age in Bangladesh with MAM. The study will be conducted in the Mirpur area within the Dhaka city. The Mirpur study/surveillance area is well known to all staff working in the Mirpur field clinic as they have been working in this area on existing studies for the last 10 years. The investigators have established a field clinic/lab located within ward 5 where staff have been working for the BEAN project (PR-14110 and PR-18036) for the last 7 years. Existing staff will therefore recruit the children and mothers from the study area. The Mirpur area is a densely populated area and is located around 8 km from the main campus of icddr, b at Mohakhali, Dhaka. Mirpur was selected as the study site because it is inhabited by poor and middle-class families, residential and sanitary conditions are typical of any congested urban settlements, and there have been ongoing research activities in this area for the last 30 years.

This study design will adequately assess the capabilities of the EF/ER Toolkit in the control group allowing comparisons to high-income country data. Through the two interventional arms, and the comparison to 3y old untreated children, there will be high quality pilot data on the EF/ER response to interventions to power a definitive trial. The enrolled children will have follow-up visits at 2 years and 3 years of age with EF/ER for developmental assessment.

ELIGIBILITY:
Inclusion criteria:

Inclusion criteria for malnourished (MAM) children at 1 and 3 years of age: All of the following criteria must be met for a subject to be eligible to participate in the study

* Mother willing to sign consent form
* Child age 12-15 months or 36-39 months of age
* WHZ <-2 and ≥-3 z-score, and/or MUAC <12.5 and ≥11.5 cm and free from any acute illness
* Mother agrees to feed their children a study diet at home.
* Mother willing to bring the child to the clinic for assessment (morbidity, nutrition history, adherence to treatment, anthropometry and advice to mother on parenting) and clinical examination.
* Mother will agree to provide her biological samples
* Mother willing to have a child undergo biological sample collection and neuropsychological assessment at baseline (1-year-old) and at ages 2 years and 3 years at the clinic.
* Family has no plan to move from the study area in the next three years.

Inclusion criteria for Control group with normal health (normal Z score):

* Mother willing to sign consent form
* Child age 12-15 months
* WHZ score > -1 and free from any acute illness
* Mother willing to bring the child to the clinic for assessment (morbidity, nutrition history, adherence to treatment, anthropometry and advice to mother on parenting) and clinical examination.
* Mother will agree to provide her biological samples (see below).
* Mother willing to have a child undergo biological sample collection and neuropsychological assessment at baseline at 1 year old and again at 2 years and 3 years at the clinic.
* Family has no plan to move from the study area in the next two years.

Exclusion Criteria:

Exclusion criteria for malnourished (MAM) children: Meeting any of the following criteria will exclude a subject from study participation

* Mother who is not willing to sign a consent form.
* Congenital anomaly.
* Mother who is not willing to feed the rehabilitation feed or the small quantity supplement to her child.
* Family will not stay 3 years in the study area.

Exclusion criteria for Control group with normal health (normal Z score): Meeting any of the following criteria will exclude a subject from study participation -

* Mother who is not willing to sign a consent form.
* Child age >15 months or < 12m.
* Mother who is not willing to feed the rehabilitation feed or the small quantity supplement to her child.
* Family will not stay 3 years in the study area.
* Any congenital anomaly.

Ages: 12 Months to 39 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 280 (Estimated)
Dates: Start 2022-02-07 (Actual); Primary Completion 2024-08 (Estimated); Study Completion 2024-08 (Estimated)

PRIMARY OUTCOMES:
Change in BAYLEY-4 scores from 1 year to 2 years of age | All enrolled children at 1 year ±1m(11m-13m) and 2 years ±1m(23m-25m)
  Bayley-4 Scales of Infant and Toddler Development is standardized developmental assessment tool for determining a child's developmental status at a given age (up to 42 months) BAYLEY-4 assess development in children of 1-42 months old in 5 domains: cognition, motor, language, socio-emotional, and adaptive behavior.

SECONDARY OUTCOMES:
Change in functional Near Infrared spectroscopy (fNIRS) from 1 year to 2 years of age | All enrolled children at 1 year ±1m(11m-13m) and 2 years ±1m(23m-25m)
  Brain activity will be assessed using fNIRS, a method that measures changes in blood oxygen concentration as a consequence of neural activity in the brain. fNIRS can be used to measure brain activity that is related to an externally presented stimulus, or it can measure the connections between brain activity in different parts of the brain with no explicit external stimulus presentation. Measures of hemodynamics reported by fNIRS include relative concentration changes in oxy-hemoglobin, deoxy-hemoglobin and total hemoglobin. The fNIRS measurement is completely non-invasive and has been used in infant studies of brain activity for over 15 years.
Change in Electroencephalogram (EEG) power from 1 year to 2 years of age | All enrolled children at 1 year ±1m(11m-13m) and 2 years ±1m(23m-25m)
  The EEG will be used to investigate functional connectivity and power spectra across different scalp regions during both rest (baseline) and task activity. In addition, we will deploy a number of perceptual and cognitive tasks while recording the event-related potential (a subset of the EEG). . ERPs measure changes in electrical activity of the brain in response to stimulus presentation (auditory, visual, etc0. In addition, sophisticated signal processing/machine learning approaches can be applied to examine EEG frequency information (e.g., theta activity, phase amplitude coupling), which could serve as indices of local circuit connectivity. The EEG works by detecting small charges emitted by the brain during activity, amplifying the signals, and graphing signals in real time.
Change in LENA (Language Environment Analysis) from 1 year to 2 years of age | Baseline at 1 year ±1m(11m-13m) for control and intervention and 3 years ±2m(34m-38m) for the outcome reference group, and during follow up of control and intervention group at 2 years ±1m(23m-25m) and 3 years ±2m(34m-38m) of age.
  The LENA recorder and software measure the frequency of vocalization/verbalizations and conversational turns in children. Digital audio recordings are collected in a participant's home at baseline visit and annually afterwards. Thus, we will be able to see the influence of language input at different crucial points in early development. Recording data at multiple time points also gives us a measure of the consistency of the language environment.
Change in Parent-Child Interaction coded data from 1 year to 2 years of age | All enrolled children at 1 year ±1m(11m-13m) and 2 years ±1m(23m-25m)
  A 10-15 minute interaction between parent and child will be recorded. Parents will be asked to engage their child in play or conversations in the presence and absence of toys and books. The child will also play with the toys/books while the parent completes short surveys or watches a short video. The interaction will be filmed and transcribed. Language transcripts and videos will be coded for the child's and parent's use of language and mutual engagement.
Change in weight in kilograms at the start of intervention until they reach within 1 standard deviation of the mean | Baseline, weekly, quarterly
  Weight will be measured at enrollment, then weekly during rehabilitation to achieve anthropometric recovery, and then quarterly for the duration of the study (till 36months of age) from 140 children who have enrolled with MAM. Weight data will also be collected from 70 normal children at enrolment, then monthly for 3 months, then quarterly for the duration of the study (until 36months of age).
Change in height in meters at the start of intervention until they reach within 1 standard deviation of the mean | Baseline, weekly, quarterly
  Height will be measured at enrollment, then weekly during rehabilitation to achieve anthropometric recovery, and then quarterly for the duration of the study (till 36months of age) from 140 children who have enrolled with MAM. Height data will also be collected from 70 normal children at enrolment, then monthly for 3 months, then quarterly for the duration of the study (until 36 months of age).
Change in Mid-upper arm circumference (MUAC) in centimeters at the start of intervention until they reach within 1 standard deviation of the mean | Baseline, weekly, quarterly
  MUAC will be measured at enrollment, then weekly during rehabilitation to achieve anthropometric recovery, and then quarterly for the duration of the study (till 36months of age) from 140 children who have enrolled with MAM. MUAC data will also be collected from 70 normal children at enrolment, then monthly for 3 months, then quarterly for the duration of the study (until 36months of age).
Change in head circumference in centimeters | Baseline, 2 years, 3 years
  Head circumference will be measured at enrollment, at the age of 2 years and 3 years.
Change in blood analytes | Baseline, 3 months, 24 months, 36 months
  2-3 ml of child blood will be collected at enrollment, at the time of achieved ideal wt/ht (anthropometry recovery) or at the end of 3 months of E-RUSF/RUSF intervention, 24 months and 36 months of age to perform concentration of 24 vitamins and mineral micro nutrients, functional lipid concentrations in red cell membrane, serum siallylated milk oligo saccharides, Lutein/ zeaxantnine / cryptoxanthine and Microbiome directed blood metabolome.
Change in stool metabolome | Baseline, 3 months, 24 months, 36 months
  Stool sample will be collected at enrollment, at the time of achieved ideal wt/ht (anthropometry recovery), or at the end of 3 months of E-RUSF/RUSF intervention, 24 months and 36 months of age to perform 16S microbial sequencing, Functional pathway analysis and stool metabolome.

CONTACTS AND LOCATIONS:
Overall Officials: Charles Nelson, Ph.D, Principal Investigator — Children's Hospital Boston/Harvard University; Terrence Forrester, Dr, Principal Investigator — University of the West Indies
Locations (1):
- International Centre for Diarrheal Disease Research, Dhaka, Bangladesh

IPD SHARING:
Plan to Share IPD: Yes
Participants will sign a form, to give us permission to release participant data information to authorized researchers and the safety committees, icddr,b Ethical Review Committee, regulatory authorities (both in Bangladesh and the United States), the study sponsor, Synapse (a research data sharing and collaboration platform) designees, and other research organizations.
Time Frame: At the end of the study, all of the specimens will be stored at icddr,b for 5 years.
Access Criteria: We will keep all information collected from you and your child confidential and locked in a secure place under the responsibility of the study investigators. Data will be saved in secure servers at icddr,b and Boston Children's Hospital. Biological samples will be stored securely without identifying information at icddr,b. Neuro imaging testing will be done in private rooms, and subjects will be coded by a de-identified number. In addition, staff and researchers have completed the Course in The Protection of Human Research Subjects.

REFERENCES:
- [Background] Bhutta ZA, Berkley JA, Bandsma RHJ, Kerac M, Trehan I, Briend A. Severe childhood malnutrition. Nat Rev Dis Primers. 2017 Sep 21;3:17067. doi: 10.1038/nrdp.2017.67. PMID 28933421
- [Background] Black RE, Allen LH, Bhutta ZA, Caulfield LE, de Onis M, Ezzati M, Mathers C, Rivera J; Maternal and Child Undernutrition Study Group. Maternal and child undernutrition: global and regional exposures and health consequences. Lancet. 2008 Jan 19;371(9608):243-60. doi: 10.1016/S0140-6736(07)61690-0. No abstract available. PMID 18207566
- [Background] Collins S, Dent N, Binns P, Bahwere P, Sadler K, Hallam A. Management of severe acute malnutrition in children. Lancet. 2006 Dec 2;368(9551):1992-2000. doi: 10.1016/S0140-6736(06)69443-9. PMID 17141707
- [Background] Prado EL, Dewey KG. Nutrition and brain development in early life. Nutr Rev. 2014 Apr;72(4):267-84. doi: 10.1111/nure.12102. Epub 2014 Mar 28. PMID 24684384
- [Background] Mora JO, Herrera MG, Sellers SG, Ortiz N. Nutrition, social environment and cognitive performance of disadvantaged Colombian children at three years (1). Prog Clin Biol Res. 1981;77:403-20. No abstract available. PMID 7335695
- [Background] Super CM, Herrera MG, Mora JO. Long-term effects of food supplementation and psychosocial intervention on the physical growth of Colombian infants at risk of malnutrition. Child Dev. 1990 Feb;61(1):29-49. PMID 2307045
- [Background] Adair LS, Pollitt E. Outcome of maternal nutritional supplementation: a comprehensive review of the Bacon Chow study. Am J Clin Nutr. 1985 May;41(5):948-78. doi: 10.1093/ajcn/41.5.948. PMID 3993612
- [Background] McKay H, Sinisterra L, McKay A, Gomez H, Lloreda P. Improving cognitive ability in chronically deprived children. Science. 1978 Apr 21;200(4339):270-8. doi: 10.1126/science.635585.
- [Background] Blanton LV, Charbonneau MR, Salih T, Barratt MJ, Venkatesh S, Ilkaveya O, Subramanian S, Manary MJ, Trehan I, Jorgensen JM, Fan YM, Henrissat B, Leyn SA, Rodionov DA, Osterman AL, Maleta KM, Newgard CB, Ashorn P, Dewey KG, Gordon JI. Gut bacteria that prevent growth impairments transmitted by microbiota from malnourished children. Science. 2016 Feb 19;351(6275):10.1126/science.aad3311 aad3311. doi: 10.1126/science.aad3311. PMID 26912898
- [Background] Cerdo T, Dieguez E, Campoy C. Early nutrition and gut microbiome: interrelationship between bacterial metabolism, immune system, brain structure, and neurodevelopment. Am J Physiol Endocrinol Metab. 2019 Oct 1;317(4):E617-E630. doi: 10.1152/ajpendo.00188.2019. Epub 2019 Jul 30. PMID 31361544
- [Background] Gunston GD, Burkimsher D, Malan H, Sive AA. Reversible cerebral shrinkage in kwashiorkor: an MRI study. Arch Dis Child. 1992 Aug;67(8):1030-2. doi: 10.1136/adc.67.8.1030. PMID 1520007
- [Background] Gordon JI, Dewey KG, Mills DA, Medzhitov RM. The human gut microbiota and undernutrition. Sci Transl Med. 2012 Jun 6;4(137):137ps12. doi: 10.1126/scitranslmed.3004347. PMID 22674549
- [Background] Million M, Diallo A, Raoult D. Gut microbiota and malnutrition. Microb Pathog. 2017 May;106:127-138. doi: 10.1016/j.micpath.2016.02.003. Epub 2016 Feb 4. PMID 26853753
- [Background] Fox SE, Levitt P, Nelson CA 3rd. How the timing and quality of early experiences influence the development of brain architecture. Child Dev. 2010 Jan-Feb;81(1):28-40. doi: 10.1111/j.1467-8624.2009.01380.x. PMID 20331653
- [Background] Charbonneau MR, O'Donnell D, Blanton LV, Totten SM, Davis JC, Barratt MJ, Cheng J, Guruge J, Talcott M, Bain JR, Muehlbauer MJ, Ilkayeva O, Wu C, Struckmeyer T, Barile D, Mangani C, Jorgensen J, Fan YM, Maleta K, Dewey KG, Ashorn P, Newgard CB, Lebrilla C, Mills DA, Gordon JI. Sialylated Milk Oligosaccharides Promote Microbiota-Dependent Growth in Models of Infant Undernutrition. Cell. 2016 Feb 25;164(5):859-71. doi: 10.1016/j.cell.2016.01.024. Epub 2016 Feb 18. PMID 26898329
- [Background] Cusick SE, Georgieff MK. The Role of Nutrition in Brain Development: The Golden Opportunity of the "First 1000 Days". J Pediatr. 2016 Aug;175:16-21. doi: 10.1016/j.jpeds.2016.05.013. Epub 2016 Jun 3. No abstract available. PMID 27266965
- [Background] Obelitz-Ryom K, Bering SB, Overgaard SH, Eskildsen SF, Ringgaard S, Olesen JL, Skovgaard K, Pankratova S, Wang B, Brunse A, Heckmann AB, Rydal MP, Sangild PT, Thymann T. Bovine Milk Oligosaccharides with Sialyllactose Improves Cognition in Preterm Pigs. Nutrients. 2019 Jun 14;11(6):1335. doi: 10.3390/nu11061335. PMID 31207876
- [Background] Choudhury N, Ahmed T, Hossain MI, Mandal BN, Mothabbir G, Rahman M, Islam MM, Husain MM, Nargis M, Rahman E. Community-based management of acute malnutrition in Bangladesh: feasibility and constraints. Food Nutr Bull. 2014 Jun;35(2):277-85. doi: 10.1177/156482651403500214. PMID 25076775
- [Background] Puett C, Coates J, Alderman H, Sadler K. Quality of care for severe acute malnutrition delivered by community health workers in southern Bangladesh. Matern Child Nutr. 2013 Jan;9(1):130-42. doi: 10.1111/j.1740-8709.2012.00409.x. Epub 2012 Apr 20. PMID 22515318
- [Background] Ahmed T, Choudhury N, Hossain MI, Tangsuphoom N, Islam MM, de Pee S, Steiger G, Fuli R, Sarker SA, Parveen M, West KP Jr, Christian P. Development and acceptability testing of ready-to-use supplementary food made from locally available food ingredients in Bangladesh. BMC Pediatr. 2014 Jun 27;14:164. doi: 10.1186/1471-2431-14-164. PMID 24972632
- [Background] Manary MJ. Local production and provision of ready-to-use therapeutic food (RUTF) spread for the treatment of severe childhood malnutrition. Food Nutr Bull. 2006 Sep;27(3 Suppl):S83-9. doi: 10.1177/15648265060273S305. PMID 17076214
- [Background] Tripp K, Perrine CG, de Campos P, Knieriemen M, Hartz R, Ali F, Jefferds ME, Kupka R. Formative research for the development of a market-based home fortification programme for young children in Niger. Matern Child Nutr. 2011 Oct;7 Suppl 3(Suppl 3):82-95. doi: 10.1111/j.1740-8709.2011.00352.x. PMID 21929637
- [Background] Paul KH, Muti M, Chasekwa B, Mbuya MN, Madzima RC, Humphrey JH, Stoltzfus RJ. Complementary feeding messages that target cultural barriers enhance both the use of lipid-based nutrient supplements and underlying feeding practices to improve infant diets in rural Zimbabwe. Matern Child Nutr. 2012 Apr;8(2):225-38. doi: 10.1111/j.1740-8709.2010.00265.x. Epub 2010 Aug 4. PMID 22405701
- [Background] Phuka J, Ashorn U, Ashorn P, Zeilani M, Cheung YB, Dewey KG, Manary M, Maleta K. Acceptability of three novel lipid-based nutrient supplements among Malawian infants and their caregivers. Matern Child Nutr. 2011 Oct;7(4):368-77. doi: 10.1111/j.1740-8709.2011.00297.x. Epub 2011 Apr 21. PMID 21518250
- [Background] Na M, Aguayo VM, Arimond M, Stewart CP. Risk factors of poor complementary feeding practices in Pakistani children aged 6-23 months: A multilevel analysis of the Demographic and Health Survey 2012-2013. Matern Child Nutr. 2017 Oct;13 Suppl 2(Suppl 2):e12463. doi: 10.1111/mcn.12463. PMID 29032630
- [Background] Wilson B, Whelan K. Prebiotic inulin-type fructans and galacto-oligosaccharides: definition, specificity, function, and application in gastrointestinal disorders. J Gastroenterol Hepatol. 2017 Mar;32 Suppl 1:64-68. doi: 10.1111/jgh.13700. PMID 28244671
- [Background] Healey G, Murphy R, Butts C, Brough L, Whelan K, Coad J. Habitual dietary fibre intake influences gut microbiota response to an inulin-type fructan prebiotic: a randomised, double-blind, placebo-controlled, cross-over, human intervention study. Br J Nutr. 2018 Jan;119(2):176-189. doi: 10.1017/S0007114517003440. Epub 2018 Jan 8. PMID 29307330
- [Background] Melendez-Martinez AJ, Mandic AI, Bantis F, Bohm V, Borge GIA, Brncic M, Bysted A, Cano MP, Dias MG, Elgersma A, Fikselova M, Garcia-Alonso J, Giuffrida D, Goncalves VSS, Hornero-Mendez D, Kljak K, Lavelli V, Manganaris GA, Mapelli-Brahm P, Marounek M, Olmedilla-Alonso B, Periago-Caston MJ, Pintea A, Sheehan JJ, Tumbas Saponjac V, Valsikova-Frey M, Meulebroek LV, O'Brien N. A comprehensive review on carotenoids in foods and feeds: status quo, applications, patents, and research needs. Crit Rev Food Sci Nutr. 2022;62(8):1999-2049. doi: 10.1080/10408398.2020.1867959. Epub 2021 Jan 5. PMID 33399015
- [Background] Grantham-McGregor S. A review of studies of the effect of severe malnutrition on mental development. J Nutr. 1995 Aug;125(8 Suppl):2233S-2238S. doi: 10.1093/jn/125.suppl_8.2233S. PMID 7542705
- [Background] Ahmed T, Mahfuz M, Islam MM, Mondal D, Hossain MI, Ahmed AS, Tofail F, Gaffar SA, Haque R, Guerrant RL, Petri WA. The MAL-ED cohort study in Mirpur, Bangladesh. Clin Infect Dis. 2014 Nov 1;59 Suppl 4:S280-6. doi: 10.1093/cid/ciu458. PMID 25305298
- [Background] Chen RY, Mostafa I, Hibberd MC, Das S, Mahfuz M, Naila NN, Islam MM, Huq S, Alam MA, Zaman MU, Raman AS, Webber D, Zhou C, Sundaresan V, Ahsan K, Meier MF, Barratt MJ, Ahmed T, Gordon JI. A Microbiota-Directed Food Intervention for Undernourished Children. N Engl J Med. 2021 Apr 22;384(16):1517-1528. doi: 10.1056/NEJMoa2023294. Epub 2021 Apr 7. PMID 33826814
- [Background] Nahar B, Hamadani JD, Ahmed T, Tofail F, Rahman A, Huda SN, Grantham-McGregor SM. Effects of psychosocial stimulation on growth and development of severely malnourished children in a nutrition unit in Bangladesh. Eur J Clin Nutr. 2009 Jun;63(6):725-31. doi: 10.1038/ejcn.2008.44. Epub 2008 Sep 3. PMID 18772893
- [Background] Perner J, Lang B. Development of theory of mind and executive control. Trends Cogn Sci. 1999 Sep;3(9):337-344. doi: 10.1016/s1364-6613(99)01362-5. PMID 10461196
- [Background] Meek JH, Firbank M, Elwell CE, Atkinson J, Braddick O, Wyatt JS. Regional hemodynamic responses to visual stimulation in awake infants. Pediatr Res. 1998 Jun;43(6):840-3. doi: 10.1203/00006450-199806000-00019. PMID 9621996
- [Background] Lloyd-Fox S, Papademetriou M, Darboe MK, Everdell NL, Wegmuller R, Prentice AM, Moore SE, Elwell CE. Functional near infrared spectroscopy (fNIRS) to assess cognitive function in infants in rural Africa. Sci Rep. 2014 Apr 22;4:4740. doi: 10.1038/srep04740. PMID 24751935
- [Background] Sideridis G, Simos P, Papanicolaou A, Fletcher J. Using Structural Equation Modeling to Assess Functional Connectivity in the Brain: Power and Sample Size Considerations. Educ Psychol Meas. 2014 Oct;74(5):733-758. doi: 10.1177/0013164414525397. PMID 25435589
- [Background] Bentler PM. Comparative fit indexes in structural models. Psychol Bull. 1990 Mar;107(2):238-46. doi: 10.1037/0033-2909.107.2.238. PMID 2320703